CLINICAL TRIAL: NCT04936776
Title: Pediatric Vaccinations
Status: Enrolling by invitation | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI- Pediatric Vaccinations
Record Dates: First submitted 2021-03-05; First posted 2021-06-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pediatric ALL; Vaccination; Immunization
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Text message 1: Text messaging frame = safety and cleanness of clinic site. Text parents of children 0-2 years old who are due and due soon for a vaccine across the entire NYU-Brooklyn Family Health Center network.
  Interventions: Behavioral: Text messaging
- Text message 2: Text messaging frame = importance of vaccines. Text parents of children 0-2 years old who are due and due soon for a vaccine across the entire NYU-Brooklyn Family Health Center network.
  Interventions: Behavioral: Text messaging
- No text message: No text sent.

INTERVENTIONS:
Behavioral: Text messaging — Text parents of children (age 0-2yrs) who are due and due soon for a vaccine across the entire NYU-Brooklyn FHC network to increase vaccination rates.
  Groups: Text message 1; Text message 2

SUMMARY:
As the Covid-19 pandemic hit New York City in the spring of 2020, many families were home-bound due to the city-wide lockdown. As a result, families in New York City were unable to attend their child's healthcare appointments and many young children did not receive their regularly-scheduled vaccinations. Parts of the city-wide lockdown did eventually lift in the summer of 2020 as positive Covid-19 virus rates declined in NYC. However, regularly scheduled vaccination rates (non-Covid-related) remain low. Yet, it is critical that young children receive their mandatory vaccines in a timely manner to decrease the chance of contracting preventable illnesses. Thus, the investigators seek to increase vaccination rates among children ages 0-2 years in Sunset Park Brooklyn.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 0-2 years with delayed vaccinations (due for vaccine and due soon) in NYU Brooklyn Family Health Centers network.

Exclusion Criteria:

* Children above the age of 2 who do not attend NYU Brooklyn Family Health Centers network

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 0-2 years with delayed vaccinations (due for vaccine and due soon) in NYU Brooklyn Family Health Centers network.
Sampling Method: Probability Sample
Enrollment: 1203 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in pediatric vaccination rate among children ages 0-2 years (proportion of vaccines due per person) | Baseline - 1 year

SECONDARY OUTCOMES:
Number of scheduled appointments | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Holly Krelle, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No